CLINICAL TRIAL: NCT00957008
Title: Use of Electronic Feedback on Diet and Physical Activity to Enhance Weight Management
Brief Title: Lifestyle Education for Activity and Nutrition for a Leaner You
Acronym: LEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Steven N. Blair, Distinguished Professor Emeritus, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00005091
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Results first posted 2011-03-23 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Body Weight Changes; Overweight
MeSH Terms: conditions — Body Weight Changes; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A - GWL (Experimental): Group Weight Loss Program (GWL) - Participants in this group attended a 14-session group weight loss program administered by trained facilitators plus 6 one-on-one telephone sessions with a facilitator.
  Interventions: Behavioral: Group weight loss program
- B - GWL+SWA (Experimental): Group weight loss program plus use of the Senseware Armband - Participants in this group attended a 14-session group weight loss program administered by trained facilitators plus 6 one-on-one telephone sessions with a facilitator and wore a SenseWear Armband. The SenseWear system includes the Armband, a real-time display device, and a personalized Weight Management Solutions web account. Participants received training in using the Armband and were asked to wear it at least 16 hours per day.
  Interventions: Other: Group weight loss program plus use of the Senseware Armband
- C - SWA Alone (Experimental): Use of the senseware armband alone program - The intervention for the SWA Alone group was the SenseWear system includes the Armband, a real-time display device, and a personalized Weight Management Solutions web account. Participants received training in using the Armband and were asked to wear it at least 16 hours per day.
  Interventions: Device: Use of the senseware armband alone program
- D - Standard Care (No Intervention): Standard Care - Participants in this group received a self-directed weight loss manual that focused on cognitive and behavior change principles and learning activities based on Active Living Every Day and Healthy Eating Every Day

INTERVENTIONS:
Behavioral: Group weight loss program — Participants will be asked to attend 14 one-and-half-hour group sessions at the University of South Carolina's Public Health Research Center (PHRC) over a 16 week period. After the groups end, they will be asked to take part in 6 telephone calls during their remaining 2 months in the program. They will also receive a weight loss manual.
  Other Names: Standard bahavior weight loss
  Arms: A - GWL
Other: Group weight loss program plus use of the Senseware Armband — Participants will be asked to attend 15 one-and-half-hour group sessions at the University of South Carolina's Public Health Research Center (PHRC) over a 17 week period. After the groups end, they will be asked to take part in 6 telephone calls during their remaining 2 months in the program. They will also receive a SenseWear Armband to wear during their 6 months in the program. One of these group sessions will be devoted to learning how to use the SenseWear Armband. They will be asked to wear the Armband regularly, upload data from the Armband to a web-based application, and input nutritional and health information into a personalized web account. They will receive a weight loss manual in addition to the group sessions and Armband.
  Other Names: Standard behavioral weight loss plus Armband
  Arms: B - GWL+SWA
Device: Use of the senseware armband alone program — Participants will be asked to attend a one-hour group session at the University of South Carolina's Public Health Research Center (PHRC) to learn how to use the SenseWear Armband. They will then be asked to take part in a follow-up telephone call one week after they start wearing the armband. For the 6 months they are in the program, they will be asked to wear the Armband regularly, upload data from the Armband to a web-based application, and input nutritional and health information into a personalized web account. They will also receive a weight loss manual in addition to the Armband.
  Other Names: Armband Alone
  Arms: C - SWA Alone

SUMMARY:
Although weight loss programs are effective in the short-term, maintaining weight loss is more challenging. Regularly tracking and logging physical activity (PA) and diet is related to greater improvements in PA and diet and to greater weight loss over time. Receiving continuous real-time feedback regarding calories burned and calories consumed could enhance weight loss maintenance. This study will examine whether a device that provides such feedback, called the SenseWear armband, enhances weight maintenance.

200 overweight adults aged 18 to 65 years will be randomly assigned to one of four groups: (1) a standard behavior change weight loss group-based program (14 group sessions over a 4 month period followed by 6 phone calls over a 5 month period), (2) a standard behavior change weight loss group-based program (15 group session over a 4 month period followed by 6 phone calls over a 5 month period) combined with the armband, (3) the armband alone (training in the use of the armband and a follow up telephone call), or (4) a self-directed weight loss control group.

Participants will be recruited through USC through listserv emails, flyers, and worksite advertisements. Interested individuals will take part in a telephone screen, an orientation, a run-in visit (which includes 2 weeks of PA and dietary logging), a baseline assessment, and a randomization visit. The intervention will then take place over a 9-month period with eligible participants. Participants will take part in follow-up assessments at month 4 and 9. Assessments at all three times will include questionnaires assessing diet, PA, psychosocial factors related to diet and PA, and quality of life related measures. They will also have their fasting blood drawn to assess lipids, glucose, and insulin, and staff will measure their blood pressure, waist circumference (size), skinfold, height, and weight.

DETAILED DESCRIPTION:
Use of Electronic Feedback on Diet and Physical Activity to Enhance Weight Management Research Summary Steven N. Blair, PED, Principal Investigator

Primary Aim

Dr. Blair and the investigative team will evaluate the contribution of the BodyMedia metabolic monitoring system to weight loss within the context of a standard behavioral weight loss program, and also as a stand alone system. The BodyMedia system consists of a metabolic monitor (armband) and computer software that analyzes energy expenditure, duration and level of physical activity, and other metabolic processes in free-living conditions. The proposed study will test the following hypotheses:

1. The standard behavioral weight loss program (Standard), BodyMedia augmented program (Armband), and the Armband Alone will produce more weight loss and reduction in waist circumference over 4 months and maintain greater weight loss and reduction in waist circumference than does a usual care self-help program (Usual Care).
2. The Armband program will produce weight loss and reduction in waist circumference comparable to the Standard program over 4 months.
3. The Armband Alone program will produce weight loss and reduction in waist circumference comparable to the Standard program after 9 months.
4. The Armband program will produce weight loss and reduction in waist circumference greater than the Standard program after 9 months.

Primary Outcomes

1. Body weight
2. Waist circumference

Secondary Outcomes

1. Weekly energy expenditure in physical activity.
2. Weekly caloric intake.
3. Percent of participants losing ≥5% of baseline body weight.
4. Stages of Motivational Readiness for physical activity and diet changes.

Tertiary Outcomes

1. Blood pressure.
2. Fasting lipid profile.
3. Fasting blood glucose.
4. Fasting blood insulin
5. Quality of life.

Study Design

The design will be a randomized controlled trial with four arms:

1. Standard behavioral weight loss intervention program.
2. Armband (standard behavioral weight loss intervention program augmented by using the BodyMedia armband and monitoring system to reinforce and support making changes in these behaviors).
3. Armband Alone that includes a one-hour orientation at baseline on how to use the armband, with a one week follow-up telephone call to answer questions.
4. Usual care (self-help with a diet and physical activity manual that provides guidance on changing these behaviors).

Fifty participants will be assigned to each of the study arms. The Standard and Armband groups will participate in weekly group counseling sessions for four months. During months 5-7 study staff will contact participants weekly via email or telephone to monitor their reports of dietary and physical activity logging, and to provide counseling support as necessary. During months 8 and 9, these contacts will be monthly. For the Armband Alone group, study staff will make monthly contact by telephone or email to answer questions and provide encouragement.

Data collection for outcomes will occur at baseline, 4 months (no blood chemistry analyses will be performed at 4 months), and 9 months. Participants will be recruited into the study over several months, and all participants will have completed the follow-up (month 9) data collection by the end of the 18-month study period.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years older men & women
* Body mass index 25.0-39.9
* Ability to provide informed consent

Exclusion Criteria:

* Type I Diabetes
* Type II diabetes taking insulin
* Surgery or Hospitalization in last year (unless minor outpatient surgery)
* Blood pressure >159/94
* Cancer (other than non-melanoma skin cancer) in last 5 years
* History of bariatric surgery
* Current treatment with herbal, over-the-counter, or prescription weight loss drugs
* Current treatment with ant-metabolite medications or other medications that affect weight
* Current pregnancy or breastfeeding, or plans pregnancy in next 18 months gastrointestinal disorders including ulcerative colitis, Crohn's disease, malabsorption syndromes)
* Chronic renal insufficiency
* Chronic liver disease
* History of anorexia nervosa, bulimia, laxative abuse
* Current alcohol or substance abuse
* Chronic heart failure, New York Heart Association Class III or IV
* Uncontrolled arrythmia
* Uncontrolled hyper- or hypothyroidism
* Large weight loss of 20 or more kilograms in the past year
* Hospitalization for mental illness within the past 5 years or currently undergoing treatment for severe mental illness
* Center for Epidemiologic Studies Depression Scale Score ≥ 16
* Musculoskeletal problems interfering with exercise.
* Autoimmune or collagen vascular diseases.
* Immunodeficiency diseases or a positive Human immunodeficiency virus test
* Unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven N Blair, PED, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina Department of Exercise Science, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Shuger SL, Barry VW, Sui X, McClain A, Hand GA, Wilcox S, Meriwether RA, Hardin JW, Blair SN. Electronic feedback in a diet- and physical activity-based lifestyle intervention for weight loss: a randomized controlled trial. Int J Behav Nutr Phys Act. 2011 May 18;8:41. doi: 10.1186/1479-5868-8-41. PMID 21592351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We conducted a total of 787 telephone screening interviews between February 2008 and February 2009 from the greater Columbia, South Carolina area. 197 men and women were eligible. Participants were recruited using a wide variety of techniques, including newspaper, mailers, community events, and worksite and other e-mail distributions.
Pre-assignment Details: Exclusion criteria included significant weight loss (>20 lbs) in the last 6 months, elevated blood pressure (160/95 mm Hg), ailments that limited their physical activity, or serious medical conditions or other issues (e.g. pregnancy or depression) contraindicating or confounding the weight loss intervention.
Groups:
- Group-based Behavioral Weight Loss Education Group (GWL): During the first 4 months of the intervention, these participants received 14 GWL sessions based on ALED and HEED. Each session followed the ALED and HEED curriculum format with the addition of a weekly weigh-in and greater emphasis on weight loss than in the original programs. During the final 5 months participants received 6 one-on-one telephone counseling sessions to provide continued support and enhance weight loss maintenance.
- Combined GWL and SWA Group (GWL+SWA): These participants received all components of the GWL including the 6 one-on-one telephone counseling sessions and also received the SenseWearTM platform.
- Armband Alone Group (SWA-alone): The SWA-alone group received the SenseWearTM platform consisting of the armband, a real-time wrist watch display, and access to a personalized Weight Management Solutions web account. While wearing the armband, participants received real-time feedback from the wrist watch on several outcomes (i.e. energy expenditure, minutes spent in moderate and vigorous physical activity, and steps per day). Feedback regarding energy balance was received as participants regularly uploaded their armband to the website and recorded daily energy intake and body weight to the Weight Management Solutions web account. Participants were asked to wear the armband 16 hours a day, 7 days a week.
- Standard Care (Control Group): Standard care participants received a self-directed weight loss manual based on two evidence-based programs, Active Living Every Day (ALED) and Healthy Eating Every Day (HEED). The manual's focus was to help individuals adopt a healthful eating pattern and increase their physical activity levels through the use of cognitive and behavioral strategies consistent with the Transtheoretical Model and Social Cognitive Theory.
Period: Overall Study
Arm/Group | Group-based Behavioral Weight Loss Education Group (GWL) | Combined GWL and SWA Group (GWL+SWA) | Armband Alone Group (SWA-alone) | Standard Care (Control Group)
Started | 49 | 49 | 49 | 50
Completed | 28 | 37 | 32 | 26
Not Completed | 21 | 12 | 17 | 24
Not completed — Withdrawal by Subject | 13 | 10 | 12 | 16
Not completed — Lost to Follow-up | 3 | 1 | 3 | 4
Not completed — Physician Decision | 1 | 0 | 1 | 1
Not completed — Relocated; Family conflict | 4 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group-based Behavioral Weight Loss Education Group (GWL) | Combined GWL and SWA Group (GWL+SWA) | Armband Alone Group (SWA-alone) | Standard Care (Control Group) | Total
Number analyzed (Participants) | 49 | 49 | 49 | 50 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 48 | 47 | 50 | 194
  >=65 years | 0 | 1 | 2 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (12.4) | 45.7 (10.4) | 47.7 (11.6) | 47.2 (8.9) | 46.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 40 | 42 | 161
  Male | 10 | 9 | 9 | 8 | 36
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 49 | 50 | 197

OUTCOME MEASURES:

1. Primary Outcome: Waist Circumference
Description: Waist circumference was measured at the level of the umbilicus with a plastic tape measure.
Time Frame: Month 9
Measure: Least Squares Mean (Standard Error); unit: cm
Groups:
- B - GWL+SWA: Group weight loss program plus use of the Senseware Armband - Participants in this group attended a 14-session group weight loss program administered by trained facilitators plus 6 one-on-one telephone sessions with a facilitator and wore a SenseWear Armband. The SenseWear system includes the Armband, a real-time display device, and a personalized Weight Management Solutions web account. Participants received training in using the Armband and were asked to wear it at least 16 hours per day.
  Group weight loss program plus use of the Senseware Armband: Participants will be asked to attend 15 one-and-half-hour group sessions at the University of South Carolina's Public Health Research Center (PHRC) over a 17 week period. After the groups end, they will be asked to take part in 6 telephone calls during their remaining 2 months in the program. They will also receive a SenseWear Armband to wear during their 6 months in the program. One of these group sessions will be devoted to learning
Arm/Group | A - GWL | B - GWL+SWA | C - SWA Alone | D - Standard Care
Number analyzed (Participants) | 49 | 49 | 49 | 50
cm | 105.87 (2.24) | 99.27 (2.22) | 102.32 (2.23) | 102.77 (2.28)

2. Primary Outcome: Body Weight
Description: Body weight was assessed using a calibrated balance-beam scale.
Time Frame: nine month
Measure: Least Squares Mean (Standard Error); unit: Kg
Arm/Group | Group-based Behavioral Weight Loss Education Group (GWL) | Combined GWL and SWA Group (GWL+SWA) | Armband Alone Group (SWA-alone) | Standard Care (Control Group)
Number analyzed (Participants) | 49 | 49 | 49 | 50
Kg | 99.98 (3.00) | 93.73 (2.99) | 97.60 (2.99) | 101.32 (3.05)

3. Primary Outcome: Body Weight
Time Frame: 4 month
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | A - GWL | B - GWL+SWA | C - SWA Alone | D - Standard Care
Number analyzed (Participants) | 49 | 49 | 49 | 50
kg | 100.74 (2.99) | 96.83 (2.99) | 98.48 (2.97) | 101.23 (3.03)

4. Primary Outcome: Waist Circumference
Time Frame: 4 month
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | A - GWL | B - GWL+SWA | C - SWA Alone | D - Standard Care
Number analyzed (Participants) | 49 | 49 | 49 | 50
cm | 107.10 (2.23) | 102.12 (2.21) | 102.99 (2.21) | 104.69 (2.26)

5. Secondary Outcome: Blood Fasting Glucose
Time Frame: Month 9
Population: Last observation carried forward
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Group-based Behavioral Weight Loss Education Group (GWL) | Combined GWL and SWA Group (GWL+SWA) | Armband Alone Group (SWA-alone) | Standard Care (Control Group)
Number analyzed (Participants) | 44 | 39 | 41 | 40
mg/dl | -5.42 [-10.21 to -0.62] | -12.59 [-17.6 to -7.57] | -8.88 [-13.76 to -4.01] | 1.99 [-2.79 to 6.76]

ADVERSE EVENTS:
Arm/Group | Group-based Behavioral Weight Loss Education Group (GWL) | Combined GWL and SWA Group (GWL+SWA) | Armband Alone Group (SWA-alone) | Standard Care (Control Group)
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/49 | 0/50

LIMITATIONS AND CAVEATS:
Large attrition rate due to time commitment; mostly female and highly educated sample; short intervention; GWL did not perform well

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes